CLINICAL TRIAL: NCT05295706
Title: Towards Understanding the Relationship Between Meals and Blood Biomarkers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Texas A&M University (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB2020-0005F
Record Dates: First submitted 2022-02-25; First posted 2022-03-25 (Actual); Last update posted 2022-05-20 (Actual); Status verified 2021-09

CONDITIONS: Type 2 Diabetes
Keywords: Continuous glucose monitoring; Dietary habits; Counterfactual thinking
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Feeding Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in this group will complete the same measures as the control group, but will additionally be involved in a counterfactual intervention conducted by an advanced graduate student.
  Interventions: Behavioral: Counterfactual Intervention
- Control Group (No Intervention): Participants in this group will complete the same measures as the experimental group. Instead of being involved in a counterfactual intervention, participants will be asked about their intentions to complete future study components.

INTERVENTIONS:
Behavioral: Counterfactual Intervention — The intervention occurs during the third study visit. This is a counterfactual intervention, which will involve asking the subjects to think of an alternative reality that "might have been" based on the concurrency of their glucose readings and the meals they ate.
  Arms: Intervention Group

SUMMARY:
The purpose of this study is to establish the reasonableness of using food-based photo diaries and continuous glucose monitors (CGM) to engage in counterfactual thinking strategies. These strategies may improve food choices among participants diagnosed with prediabetes (intervention group).

DETAILED DESCRIPTION:
The long-term objective of this project is to create a counterfactual-based lifestyle intervention that curtails the progression of prediabetes to T2DM through management and knowledge of food choices. This is a significant objective since 70% of prediabetes patients go on to develop T2DM. The project addresses a major objective of PATHS-UP in general and Thrust 4 in particular, by developing an innovative behavior-change intervention that will eventually make use of information from the Lab-on-your-Wrist device. To our knowledge, this is the first project to (1) propose an intervention based on counterfactual thinking for diabetes prevention and (2) combine continuous glucose monitors (CGMs) and food photography to promote a better understanding of how food choices affect blood glucose.The specific aim of this project is to establish the validity of leveraging photo-based food diaries and CGMs to engage counterfactual thinking strategies that improve food choices amongst prediabetes participants. This will be measured by changes in (1) eating attitudes and behaviors, (2) behavioral intentions to improve healthy eating behavior, (3) motivation to improve eating behavior, (4) increased self- efficacy for healthy eating, and (5) number of glucose excursions and time-in-range.

ELIGIBILITY:
Inclusion Criteria:

* Ability to walk, sit down and stand up independently
* Family history of type 2 diabetes
* Overweight/obese status (BMI>= 25)
* Subject is judged to be in satisfactory health based on medical history, physical examination
* Willingness and ability to comply with the protocol
* HbA1C levels are within the pre-diabetic range (5.7-6.4%) or fasting plasma glucose 100-125 mg/dL
* Access to a smartphone device and willing to use WhatsApp to communicate with research personnel

Exclusion Criteria:

* Subject has planned elective surgery requiring 2 or more days of hospitalization during the entire study
* Planned medical procedures that are documented to interfere with CGM readings, such as:

  * Xylose absorption testing (oral sugar testing)
  * CT
  * MRI
  * X-ray
  * Diathermy treatment (high-frequency electric current to stimulate heat generation within body tissues)
* Established diagnosis of malignancy
* Presence of acute illness or metabolically unstable chronic illness
* Any other condition according to the PI, nurse, or study coordinator that was found during the screening visit, that would interfere with the study or safety of the patient
* Failure to give informed consent or Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in average daily glucose level | Data will be collected in between study visits 1-4 (at baseline, 3 weeks, 4 weeks, and 6 weeks)
  Collected via the Freestyle Libre Pro continuous glucose monitor placed on the participants' upper arm.
Change in number of glucose excursions and time in range | Data will be collected in between study visits 1-4 (at baseline, 3 weeks, 4 weeks, and 6 weeks)
  Collected via the Freestyle Libre Pro continuous glucose monitor placed on the participants' upper arm.
Change in HbA1C | A blood sample will be collected at the screening visit, and at 6 weeks (Study Visit #4), 14 weeks (Study Visit #5), and 22 weeks (Study Visit #6).
  Blood will be sampled through venipuncture technique on the upper arm. A blood sample of 4 mL will be collected for each measurement of the subject's A1c.

SECONDARY OUTCOMES:
Change in the Self Regulation of Eating Behaviors Questionnaire (SREBQ) scores | Collected via survey measures at baseline (Study Visit #1), 4 weeks (Study Visit #3), at 6 weeks (Study Visit #4), 14 weeks (Study Visit #5), and 22 weeks (Study Visit #6).
  Participants will report their ability to regulate and/or change their eating habits. Items correspond to a Likert style format ranging from 1 (never) to 5 (always), where higher scores indicate worse regulation (aside from one item that must be reverse-scored).
Change in General Health Intentions (GHI) scores | Self-report general health intentions data will be collected at baseline (Study Visit #1), 4 weeks (Study Visit #3), 6 weeks (Study Visit #4), 14 weeks (Study Visit #5), and 22 weeks (Study Visit #6).
  Participants will self-report their intentions to engage in healthier food habits over the next six months. Participants respond using a Likert scale ranging from 1 (strongly disagree) to 7 (strongly agree), where higher scores indicate greater intentions to eat healthy.
Change in Regulation of Eating Behaviors Scale (REBS) scores | Collected via survey measures at baseline (Study Visit #1), 6 weeks (Study Visit #4), 14 weeks (Study Visit #5), and 22 weeks (Study Visit #6).
  Participants will self-report their motivations for eating via the Regulation of Eating Behaviors Scale, including whether they eat to cope with negative affect, to be social, to comply with others' expectations, and to enhance pleasure. Scores are measured on a Likert scale from 1 (does not correspond at all) to 7 (corresponds exactly), where higher scores indicate greater regulation of eating behaviors (with the exception of a few items that must be reverse-scored).
Change in the Eating Self-Efficacy Scale (ESES) scores | Data will be collected at baseline (Study Visit #1), 6 weeks (Study Visit #4), 14 weeks (Study Visit #5), and 22 weeks (Study Visit #6).
  Participants respond to a survey (ESES) intended to measure self-efficacy and self-regulation of healthy eating. Items are answered using a Likert scale ranging from 1 (not difficult at all) to 7 (extremely difficult), where higher scores indicate greater use of excessive food intake in social and emotional situations.
Change in the Behavioral Strategies - Engagement and Intentions score | Collected once per week over the first 6 weeks.
  Collected via questions developed through this study (Behavioral Strategies - Engagement and Intentions) by lead investigators asking about participant's (experimental group only) use of counterfactual strategies developed during Study Visit #3 (3 weeks) (e.g., "Reduce rice intake"). Responses are answered using a Likert scale ranging from 1 (none of the time) to 7 (most of the time), where higher scores indicate greater engagement and intentions to use behavioral strategies.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Translational Research in Age and Longevity, College Station, Texas, United States

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT05295706/Prot_000.pdf
  • Informed Consent Form (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/06/NCT05295706/ICF_001.pdf